CLINICAL TRIAL: NCT00770510
Title: A Phase II/III Study of SEP-190 (Eszopiclone) in Patients With Primary Insomnia
Brief Title: A Phase II/III Study of SEP-190 (Eszopiclone) in Patients With Primary Insomnia (Study 190-126)
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Eisai Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 190-126
Record Dates: First submitted 2008-10-09; First posted 2008-10-10 (Estimated); Results first posted 2013-02-04 (Estimated); Last update posted 2013-02-04 (Estimated); Status verified 2012-12

CONDITIONS: Primary Insomnia
Keywords: Primary insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Eszopiclone; Zolpidem

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- Eszopiclone 1 mg (Experimental)
  Interventions: Drug: Eszopiclone 1 mg
- Eszopiclone 2 mg (Experimental)
  Interventions: Drug: Eszopiclone 2 mg
- Eszopiclone 3 mg (Experimental)
  Interventions: Drug: Eszopiclone 3 mg
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Zolpidem Tartrate 10 mg (Active Comparator)
  Interventions: Drug: Zolpidem Tartrate 10 mg

INTERVENTIONS:
Drug: Eszopiclone 1 mg — Eszopiclone 1 mg tablet, taken orally at bed time for 2 consecutive nights. Each participant was assigned to one of 10 prespecified treatment sequence patterns. Each interval (five total intervals) of 2 consecutive nights was separated by a washout of approximately 5 days. A follow-up period consisted of 6 days.
  Other Names: SEP-190
  Arms: Eszopiclone 1 mg
Drug: Eszopiclone 2 mg — Eszopiclone 2 mg tablet, taken orally at bed time for 2 consecutive nights. Each participant was assigned to one of 10 prespecified treatment sequence patterns. Each interval (five total intervals) of 2 consecutive nights was separated by a washout of approximately 5 days. A follow-up period consisted of 6 days.
  Other Names: SEP-190
  Arms: Eszopiclone 2 mg
Drug: Eszopiclone 3 mg — Eszopiclone 3 mg tablet, taken orally at bed time for 2 consecutive nights. Each participant was assigned to one of 10 prespecified treatment sequence patterns. Each interval (five total intervals) of 2 consecutive nights was separated by a washout of approximately 5 days. A follow-up period consisted of 6 days.
  Other Names: SEP-190
  Arms: Eszopiclone 3 mg
Drug: Placebo — Placebo tablet, taken orally at bed time for 2 consecutive nights. Each participant was assigned to one of 10 prespecified treatment sequence patterns. Each interval (five total intervals) of 2 consecutive nights was separated by a washout of approximately 5 days. A follow-up period consisted of 6 days.
  Arms: Placebo
Drug: Zolpidem Tartrate 10 mg — Zolpidem Tartrate 10 mg tablet, taken orally at bed time for 2 consecutive nights. Each participant was assigned to one of 10 prespecified treatment sequence patterns. Each interval (five total intervals) of 2 consecutive nights was separated by a washout of approximately 5 days. A follow-up period consisted of 6 days.
  Arms: Zolpidem Tartrate 10 mg

SUMMARY:
The purpose of this study is to investigate and evaluate the efficacy of Eszopiclone in Japanese participants with primary insomnia.

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind, placebo-controlled, 5-way cross-over study to investigate and evaluate the efficacy of eszopiclone in Japanese participants with primary insomnia. The treatment period consists of two consecutive days (two nights) as one term. Patients will receive oral eszopiclone (1, 2, 3 mg), zolpidem tartrate (10 mg), or placebo once daily at bedtime for each use. Participants were randomly assigned to one of 10 prespecified treatment sequence patterns.

ELIGIBILITY:
Inclusion Criteria:

1. Participants aged greater than or equal to 21 and less than 65 years at the time of obtaining written informed consent
2. Participants diagnosed with primary insomnia based on the Diagnostic and Statistical Manual of Mental Disorders, text revision (DSM-IV-TR) Japanese version and have both of the following conditions which are persistent for more than or equal to 4 weeks before the start of observation period:

   * Sleep latency of more than or equal to 30 minutes for more than or equal to 3 days a week
   * Total sleep time of less than or equal to 390 minutes for more than or equal to 3 days a week
3. Participants who meet both of the following based on polysomnogram (PSG) in observation period:

   * Objective sleep latency of more than or equal to 20 minutes for 2 consecutive PSG days
   * Objective total sleep time of less than or equal to 420 minutes for 2 consecutive PSG days, or objective wake time during sleep of more than or equal to 20 minutes for 2 consecutive PSG days

Exclusion Criteria:

1. Participants with comorbid primary sleep disorders (e.g., circadian rhythm disorder, restless limb syndrome, periodic limb movement disorder, sleep apnea syndrome), other than primary insomnia.
2. Participants with insomnia caused by pharmacological actions (drug-induced insomnia).
3. Participants with comorbid sleep disorder associated with other disease(s) such as psychiatric and/or physical disease(s).
4. Participants with a complication of psychiatric disorders in Axis I or personality disorder in Axis II defined in DSM-IV-TR Japanese version.
5. Participants with organic mental disorder.

Ages: 21 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 192 (Actual)
Dates: Start 2008-09; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Atsushi Kamijo, Study Director — New Product Development Department, Clinical Research Center
Locations (20):
- Japan (20):
  - Toyohashi, Aichi-ken
  - Akita, Akita
  - Fukuoka, Fukuoka
  - Kitakyushu, Fukuoka
  - Kurume, Fukuoka
  - Gifu, Gifu
  - Hiroshima, Hiroshima
  - Otaru, Hokkaido
  - Sapporo, Hokkaido
  - Kagoshima, Kagoshima-ken
  - Kawasaki, Kanagawa
  - Kochi, Kochi
  - Kumamoto, Kumamoto
  - Kyoto, Kyoto
  - Urazoe, Okinawa
  - Osaka, Osaka
  - Sakai, Osaka
  - Kodaira, Tokyo
  - Setagaya City, Tokyo
  - Shibuya City, Tokyo

REFERENCES:
- [Derived] Uchimura N, Kamijo A, Kuwahara H, Uchiyama M, Shimizu T, Chiba S, Inoue Y. A randomized placebo-controlled polysomnographic study of eszopiclone in Japanese patients with primary insomnia. Sleep Med. 2012 Dec;13(10):1247-53. doi: 10.1016/j.sleep.2012.08.015. Epub 2012 Oct 11. PMID 23063301

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was recruited at 21 centers in Japan.
Pre-assignment Details: Of the 192 participants who entered the screening period, 72 were randomized to study medication (excluding 119 ineligible participants; one withdrawal of consent).
Groups:
- Entire Study Population: Includes groups randomized to receive one of 10 prespecified treatment sequence patterns which included receiving: Eszopiclone 1 mg first, Eszopiclone 2 mg first, Eszopiclone 3 mg first, Placebo first, and Zolpidem Tartrate 10 mg first.
  Group 1: ABECD (n=7) Group 2: BCADE (n=7) Group 3: CDBEA (n=7) Group 4: DECAB (n=8) Group 5: EADBC (n=7) Group 6: DCEBA (n=8) Group 7: EDACB (n=7) Group 8: AEBDC (n=7) Group 9: BACED (n=7) Group 10: CBDAE (n=7)
  A= Eszopiclone 3 mg; B= Eszopiclone 2 mg; C= Eszopiclone 1mg; D= Placebo; E: Zolpidem 10 mg
Period: Overall Study
Arm/Group | Entire Study Population
Started | 72
Completed | 67
Not Completed | 5
Not completed — Lost to Follow-up | 2
Not completed — Pregnancy | 1
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Entire Study Population
Number analyzed (Participants) | 72
Age Continuous [Mean (Standard Deviation); unit: years] | 39.4 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 43

OUTCOME MEASURES:

1. Primary Outcome: Latency To Persistent Sleep (LPS)
Description: The objective measure, LPS, defined as the amount of time measured in minutes it takes to fall asleep was based on polysomnography (PSG) objective assessments of sleep disturbance. PSG recording was performed according to a manual for overnight PSG. The start time for PSG recording was individualized and scheduled within +/- 30 minutes of the participant's median bedtime as recorded in the sleep diary. During the screening period, participants were provided a diary in which they recorded the time of lights out before bedtime for 1 week pror to PSG evaluations. PSG recording duration for scoring was 8 hours. PSG data recorded during treatment were centrally scored by a trained expert.
Time Frame: 10 days (5 intervals of two consecutive nights)
Population: Full analysis set: includes randomized participants who were administered >= 1 dose of study medication and had evaluable data for the primary efficacy assessments from any of the 5 treatment intervals.
Measure: Mean (Standard Deviation); unit: Minutes
Groups:
- Placebo: Placebo tablet taken orally at bedtime for 2 consecutive nights in one of 5 cross-over intervals in each of 10 prespecified treatment sequence patterns.
- Eszopiclone 1 mg: Eszopiclone 1 mg tablet taken orally at bedtime for 2 consecutive nights in one of 5 cross-over intervals in each of 10 prespecified treatment sequence patterns.
- Eszopiclone 2 mg: Eszopiclone 2 mg tablet taken orally at bedtime for 2 consecutive nights in one of 5 cross-over intervals in each of 10 prespecified treatment sequence patterns.
- Eszopiclone 3 mg: Eszopiclone 3 mg tablet taken orally at bedtime for 2 consecutive nights in one of 5 cross-over intervals in each of 10 prespecified treatment sequence patterns.
- Zolpidem Tartrate 10 mg: Zolpidem Tartrate 10 mg tablet taken orally at bedtime for 2 consecutive nights in one of 5 cross-over intervals in each of 10 prespecified treatment sequence patterns.
Arm/Group | Placebo | Eszopiclone 1 mg | Eszopiclone 2 mg | Eszopiclone 3 mg | Zolpidem Tartrate 10 mg
Number analyzed (Participants) | 71 | 70 | 69 | 68 | 70
Minutes | 37.5 (37.8) | 24.4 (22.7) | 20.9 (24.3) | 12.8 (11.2) | 14.3 (22.6)

2. Secondary Outcome: Total Sleep Time (Objective & Subjective)
Description: Total sleep time defined as total sleeping time from bedtime to final awakening (measured in minutes) was objectively determined by polysomnography and subjectively determined based on participant-reported measures following treatment.
  The objective total sleep time was based on PSG-based assessments. PSG recording was performed according to a manual for overnight PSG. The start time for PSG recording was individualized and scheduled within +/- 30 minutes of the participant's median bedtime as recorded in the sleep diary. PSG recording duration for scoring was 8 hours. PSG data recorded during treatment were centrally scored by a trained expert.
  The subjective measure was based on participant-reported subjective assessments of sleep disturbance and were obtained from participants' responses to morning questionnaires. Questionnaires were administered during each visit during the treatment period.
Time Frame: 10 days (5 intervals of two consecutive nights)
Population: as for outcome 1
Measure: Median (Full Range); unit: Minutes
Arm/Group | Placebo | Eszopiclone 1 mg | Eszopiclone 2 mg | Eszopiclone 3 mg | Zolpidem Tartrate 10 mg
Number analyzed (Participants) | 71 | 70 | 69 | 68 | 70
Minutes
  Objective Total Sleep Time | 414.0 [279.3 to 470.3] | 438.3 [292.3 to 468.5] | 452.5 [227.5 to 475.8] | 453.4 [313.5 to 474.5] | 448.6 [338.8 to 476.3]
  Subjective Total Sleep Time | 360.0 [90.0 to 452.5] | 390.0 [225.0 to 460.0] | 397.5 [225.0 to 478.5] | 420.0 [225.0 to 480.0] | 411.3 [195.0 to 480.0]

3. Secondary Outcome: Sleep Efficiency
Description: Sleep efficiency (SE) was an assessment obtained from PSG during the treatment period and was defined as the ratio of total sleep time to the total time in bed of 8 hours * 100, expressed as a percent.
  PSG recording was performed according to a manual for overnight PSG. The start time for PSG recording was individualized and scheduled within +/- 30 minutes of the patient's median bedtime as recorded in the sleep diary. During the screening period, participants were provided a diary in which they recorded the time of lights out before bedtime for 1 week pror to PSG evaluations. PSG recording duration for scoring was 8 hours. PSG data recorded during treatment were centrally scored by a trained expert.
Time Frame: 10 days (5 intervals of two consecutive nights)
Population: as for outcome 1
Measure: Median (Full Range); unit: Percentage of time asleep of 8 hours
Arm/Group | Placebo | Eszopiclone 1 mg | Eszopiclone 2 mg | Eszopiclone 3 mg | Zolpidem Tartrate 10 mg
Number analyzed (Participants) | 71 | 70 | 69 | 68 | 70
Percentage of time asleep of 8 hours | 86.3 [58.2 to 98.0] | 91.3 [60.9 to 97.6] | 94.3 [47.4 to 99.2] | 94.5 [65.3 to 98.9] | 93.5 [70.6 to 99.3]

4. Secondary Outcome: Wake Time After Sleep Onset (WASO)- Objective & Subjective
Description: Wake Time After Sleep Onset (WASO) defined as total awakening time from falling asleep to final awakening was objectively determined by polysomnography and subjectively determined based on participant-reported measures following treatment.
  The objective WASO was based on PSG assessments. PSG recording was performed according to a manual for overnight PSG. The start time for PSG recording was individualized and scheduled within +/- 30 minutes of the participant's median bedtime as recorded in the sleep diary. PSG recording duration for scoring was 8 hours. PSG data recorded during treatment were centrally scored by a trained expert.
  The subjective measure was based on participant-reported subjective assessments and were obtained from participants' responses to morning questionnaires. Questionnaires were administered during each visit during the treatment period.
Time Frame: 10 days (5 intervals of two consecutive nights)
Population: as for outcome 1
Measure: Median (Full Range); unit: Minutes
Arm/Group | Placebo | Eszopiclone 1 mg | Eszopiclone 2 mg | Eszopiclone 3 mg | Zolpidem Tartrate 10 mg
Number analyzed (Participants) | 71 | 70 | 69 | 68 | 70
Minutes
  Objective Wake Time After Sleep Onset | 26.3 [1.5 to 164.3] | 22.5 [1.0 to 144.8] | 17.8 [0.5 to 176.0] | 18.8 [0.8 to 165.5] | 20.0 [1.5 to 139.5]
  Subjective Wake Time After Sleep Onset | 75.0 [3.0 to 300.0] | 60.0 [0.5 to 285.0] | 37.5 [0.0 to 255.0] | 40.0 [0.0 to 227.5] | 50.0 [0.0 to 285.0]

5. Secondary Outcome: Number of Awakenings (Objective & Subjective)
Description: Number of awakenings defined as the total number of spontaneous awakenings from falling asleep to final awakening was objectively determined by polysomnography and subjectively determined based on participant-reported measures following treatment.
  The objective number of awakenings was based on PSG assessments. PSG recording was performed according to a manual for overnight PSG. The start time for PSG recording was individualized and scheduled within +/- 30 minutes of the participant's median bedtime as recorded in the sleep diary. PSG recording duration for scoring was 8 hours. PSG data recorded during treatment were centrally scored by a trained expert.
  The subjective measure was based on participant-reported subjective assessments and were obtained from participants' responses to morning questionnaires. Questionnaires were administered during each visit during the treatment period.
Time Frame: 10 days (5 intervals of two consecutive nights)
Population: as for outcome 1
Measure: Median (Full Range); unit: Number of awakenings
Arm/Group | Placebo | Eszopiclone 1 mg | Eszopiclone 2 mg | Eszopiclone 3 mg | Zolpidem Tartrate 10 mg
Number analyzed (Participants) | 71 | 70 | 69 | 68 | 70
Number of awakenings
  Objective Number of Awakenings | 4.0 [0.5 to 18.0] | 4.0 [0.0 to 11.0] | 3.5 [0.0 to 10.0] | 2.8 [0.0 to 10.0] | 3.5 [0.5 to 14.0]
  Subjective Number of Awakenings | 3.0 [0.0 to 11.0] | 3.0 [0.5 to 8.0] | 2.5 [0.0 to 6.5] | 2.0 [0.0 to 8.0] | 2.0 [0.0 to 6.0]

6. Primary Outcome: Sleep Latency (SL)
Description: The subjective measure, SL, defined as the amount of time measured in minutes it takes to fall asleep was based on participant-reported subjective assessments of sleep disturbance and was obtained from participants' responses to morning questionnaires. Questionnaires were administered during each visit during the treatment period.
Time Frame: 10 days (5 intervals of two consecutive nights)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Placebo | Eszopiclone 1 mg | Eszopiclone 2 mg | Eszopiclone 3 mg | Zolpidem Tartrate 10 mg
Number analyzed (Participants) | 71 | 70 | 69 | 68 | 70
Minutes | 62.0 (47.8) | 45.5 (36.7) | 32.6 (26.4) | 28.4 (23.8) | 28.0 (24.6)

ADVERSE EVENTS:
Description: Safety population included randomized participants who were administered >= 1 dose of study medication and had any evaluable safety data.
Arm/Group | Placebo | Eszopiclone 1 mg | Eszopiclone 2 mg | Eszopiclone 3 mg | Zolpidem Tartrate 10 mg
Serious Adverse Events (participants affected / at risk) | 0/71 | 0/70 | 0/69 | 0/68 | 0/70
Other Adverse Events (participants affected / at risk) | 5/71 | 10/70 | 10/69 | 17/68 | 8/70
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=71) | Eszopiclone 1 mg (N=70) | Eszopiclone 2 mg (N=69) | Eszopiclone 3 mg (N=68) | Zolpidem Tartrate 10 mg (N=70)
Dysgeusia (Nervous system disorders) | 1 | 4 | 6 | 11 | 1
Somnolence (Nervous system disorders) | 2 | 1 | 3 | 4 | 3
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 2 | 3
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 2 | 2 | 1 | 0 | 1
Feeling Abnormal (General disorders) | 0 | 3 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No